CLINICAL TRIAL: NCT03522727
Title: Using Implementation Intentions to Self-incentivise Weight-loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manchester (Other)
Responsible Party: Principal Investigator, Christopher Armitage, Professor of Health Psychology, University of Manchester
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Davids/Coulthard_1
Record Dates: First submitted 2018-05-01; First posted 2018-05-11 (Actual); Last update posted 2018-10-23 (Actual); Status verified 2018-10

CONDITIONS: Overweight
MeSH Terms: conditions — Overweight

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (No Intervention): Participants will be asked to complete a questionnaire.
- Intervention 1 (Experimental): Single self-incentivising implementation intention
  After completing a questionnaire, participants will be asked to form a self-incentivising implementation intention:
  Research shows that rewarding yourself for success can help you to lose weight, but that people often forget to reward themselves. We want you to plan to reward yourself if you achieve your personal weight-loss goal, at the end of 4 weeks. To help you do this, we would like you to complete the following sentence by telling us how you will reward yourself.
  Please complete the following sentence with a reward of your own choosing.
  If I lose at least ___lbs/kg by the end of 4 weeks, then I will reward myself by…
  **Drop down menu**
  Learning a new skill...
  Interventions: Behavioral: Single self-incentivising implementation intention
- Intervention 2 (Experimental): Multiple self-incentivising implementation intentions
  After completing a questionnaire, participants will be asked to form self-incentivising implementation intentions:
  Research shows that rewarding yourself for success can help you to lose weight, but that people often forget to reward themselves. We want you to plan to reward yourself if you achieve your personal weight-loss goal, at the end of 4 weeks. To help you do this, we would like you to complete the following sentence by telling us how you will reward yourself. You can choose as many rewards as you like! Please complete the following sentence with a reward of your own choosing.
  If I lose at least ___lbs/kg by the end of 4 weeks, then I will reward myself by… and/or…
  **Drop down menu**
  Learning a new skill...
  Interventions: Behavioral: Multiple self-incentivising implementation intentions
- Intervention 3 (Experimental): Self-generated self-incentivising implementation intentions
  After completing a questionnaire, participants will be asked to form a self-incentivising implementation intention:
  Research shows that rewarding yourself for success can help you to lose weight, but that people often forget to reward themselves. We want you to plan to reward yourself if you achieve your personal weight-loss goal, at the end of 4 weeks. To help you do this, we would like you to complete the following sentence by telling us how you will reward yourself.
  Please complete the following sentence with a reward of your own choosing.
  If I lose at least ___lbs/kg by the end of 4 weeks, then I will reward myself by…
  Interventions: Behavioral: Self-generated self-incentivising implementation intentions

INTERVENTIONS:
Behavioral: Single self-incentivising implementation intention — Participants are asked to form a single self-incentivising implementation intention (if-then plans)
  Arms: Intervention 1
Behavioral: Multiple self-incentivising implementation intentions — Participants are asked to form multiple self-incentivising implementation intentions (if-then plans)
  Arms: Intervention 2
Behavioral: Self-generated self-incentivising implementation intentions — Participants are asked to form a self-incentivising implementation intention (if-then plans) without a drop-down menu
  Arms: Intervention 3

SUMMARY:
The aim of the present research is to test the effect of helping people to reward themselves when they have successfully lost weight and the impact this will have on subsequent weight. Each participant will be randomly allocated to one of four conditions. The trial requires 200 participants to perform a fully powered statistical analysis. The four conditions are: (1) a control condition, (2) intervention 1 (form a single self-incentivising implementation intention from a drop-down menu), (3) intervention 2 (form multiple self-incentivising implementation intentions from a drop-down menu), or (4) intervention 3 (asked to form a single self-incentivising implementation intention of their own devising). The main outcome measure will be BMI, which will be self-reported.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18+

Exclusion Criteria:

* Unable or unwilling to complete questionnaire

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2018-05-04 (Actual); Primary Completion 2018-07-25 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Body Mass Index | 4 weeks
  Self-reported
Actual Use of Self-Rewards | 4 weeks
  Self-reported

SECONDARY OUTCOMES:
Capabilities, opportunities and motivations | 4 weeks
  Self-reported

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Armitage, PhD, Principal Investigator — University of Manchester
Locations (2):
- United Kingdom (2):
  - Online study, Manchester
  - University of Manchester, Manchester